CLINICAL TRIAL: NCT01036282
Title: Computerized Cognitive Skills Training in Severe Mental Illness
Brief Title: Cognitive Skills Training Using Computer for Patients With Severe Mental Illness
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nathan Kline Institute for Psychiatric Research (Other)
Collaborators: Manhattan Psychiatric Center (Other)
Responsible Party: Principal Investigator, Jean-Pierre Lindenmayer, Director of Research, Nathan Kline Institute for Psychiatric Research
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 03I/C14
Record Dates: First submitted 2009-12-18; First posted 2009-12-21 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: Two arm, parallel group, randomized, blinded 12 -week intervention study of two forms of cognitive remediation in patients with chronic schizophrenia
Who Masked: Outcomes Assessor
Masking Description: Raters were blind to the type of interventions
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Computerized Cognitive Remediation (Experimental): Two arms: 1. Computerized Cognitive Remediation treatment using COGPACK. and 2. PositScience. Each arm is further randomized to either MindReader or no Mindreader.(Social Cognition Training).
  Interventions: Behavioral: Computerized Cognitive Skill Training
- CRT + Social Cognition Training (Experimental): Two 45-minute sessions of Computerized Cognitive Remediation using COGPACK, one 45-minute discussion session, plus one 45 minute Mind Reader Interactive Guide to Emotions per week for 12 weeks. compared to two 45-minute sessions of PositScience, plus one 45-min Discussion session plus one minute of Mind Reader, Interactive Guide to Emotions
  Interventions: Behavioral: CRT and Social Cognition

INTERVENTIONS:
Behavioral: Computerized Cognitive Skill Training — Behavioral: Cognitive Remediation 45 mins 2 times per week sessions of cognitive remediation (COGPACK) over twelve weeks.
  Other Names: Cognitive Remediation Therapy
  Arms: Computerized Cognitive Remediation
Behavioral: CRT and Social Cognition — Mind Reading, The Interactive Guide to Emotions for one 45 minute session per week for 12 weeks.
  Other Names: Social Emotional Functioning
  Arms: CRT + Social Cognition Training

SUMMARY:
The study is designed to evaluate the effectiveness of computerized cognitive skills training for improving memory and problem-solving skills in inpatients with schizophrenia.

DETAILED DESCRIPTION:
Subjects are stable inpatients and outpatients with schizophrenia or schizoaffective disorder who are receiving atipsychotic medication at Manhattan Psychiatric Center.

Patients receive baseline assessments (MCCB-MATRICS; Personal and Social Performance Scale, FEDT/FEIT and PANSS) and then are assigned to Cognitive Remediation (CRT) using the COGPACK program, patients are then randomly assigned to a social cognition program (Mind Reader Interactive Guide to Emotions) for a period of 12 weeks. Following 12 weeks of treatment in either CRT + Mind Reader or CRT alone, assessments are repeated by raters.

Cognitive Remediation (CRT): CRT (COGPACK, Marker and Olbrich, 1998) consists of computerized practice tests for seven cognitive domains. There are 64 programs for testing and training, each with several variants for the domains of visuomotor skills, comprehension, reaction, vigilance, memory, language, and intellectual skills. Exercises in COGPACK can be edited and expanded. Patients attend 2 (45-minutes each) groups and 1 discussion group.

Social Cognition Training: Mind Reader (Baron-Cohen et al, 2004) is an interactive computerized program of emotions and mental states. It is based on a taxonomic system of 412 emotions and mental states, grouped into 24 emotion groups, and six developmental levels (from age 4 to adulthood). The emotions and mental states are organized systematically, according to the emotion groups and developmental levels. Patients assigned to Mind Reader attend 1 group per week.

Both the CRT and Mind Reader are administered in small groups of six to eight patients each.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and above;
2. In- and out-patients;
3. DSM-IV diagnosis of schizophrenia (all subtypes) or schizoaffective disorder with illness duration >5 years;
4. Auditory and visual acuity adequate to complete cognitive tests;
5. Stable dose of oral atypical antipsychotic for at least 4 weeks;
6. Total PANSS score > 60;
7. Good physical health determined by physical examination from medical chart review;
8. Capacity and willingness to give written informed consent.
9. MMSE > 24

Exclusion Criteria:

1. Inability to read or speak English;
2. Documented disease of the central nervous system;
3. History of intellectual impairment pre-dating onset of symptoms of psychosis (e.g. mental retardation);
4. Clinically significant or unstable cardiovascular, renal, hepatic, gastrointestinal, pulmonary or hematological conditions;
5. HIV +;
6. Patients diagnosed with substance dependence;
7. Currently participating in another experimental study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 448 (Actual)
Dates: Start 2003-02 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) | Week 0, and Week 12 (after completion of Cognitive Remediation)
  Comprehensive battery of neuro-cognitive tests

SECONDARY OUTCOMES:
Facial Emotional Discrimination Task (FEDT) and Facial Emotional Identification Task (FEIT) | Week 0, and Week 12 (after compeltion of Cognitive Remediation)
  Test of facial emotion presentations on pictures to patients
Personal and Social Performance Scale (PSP) | Week 0, and Week 12 after completion of Cognitive Remediation
  Social function scale with four sub domains of social functioning
Positive and Negative Syndrome Scale (PANSS) | Week 0, Week 6 (Midpoint) and Week 12 after completion of Cognitive Remediation
  30 item Gold standard for measurement of psychiatric symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Lindenmayer, M.D., Principal Investigator — Nathan S. Kline Institute for Psychiatric Research and Manhattan Psychiatric Center
Locations (1):
- Manhattan Psychiatric Center, New York, New York, United States

REFERENCES:
- [Result] Lindenmayer JP, McGurk SR, Mueser KT, Khan A, Wance D, Hoffman L, Wolfe R, Xie H. A randomized controlled trial of cognitive remediation among inpatients with persistent mental illness. Psychiatr Serv. 2008 Mar;59(3):241-7. doi: 10.1176/ps.2008.59.3.241. PMID 18308903
- [Derived] Lindenmayer JP, Fregenti S, Kang G, Ozog V, Ljuri I, Khan A, Goldring A, McGurk SR. The relationship of cognitive improvement after cognitive remediation with social functioning in patients with schizophrenia and severe cognitive deficits. Schizophr Res. 2017 Jul;185:154-160. doi: 10.1016/j.schres.2017.01.007. Epub 2017 Jan 13. PMID 28094171